CLINICAL TRIAL: NCT06758895
Title: Cardiac Magnetic Resonance Predictors of Outcome of Rhythm Control in Patients with Atrial Fibrillation/Flutter
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maryam Ashraf Abd El-Naeem Sayed, Resident Doctor at Assiut University Heart Hospital, Assiut University
Other Study IDs: CMR in rythm control
Record Dates: First submitted 2024-12-17; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Rhythm Monitoring
Keywords: CMR predictors of rhythm control in patient with AFibirilation/flutter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
evaluate the impact of various features in CMR on the mid-term/long-term success rate of rhythm control for paroxysmal atrial fibrillation/flutter .

DETAILED DESCRIPTION:
* Atrial fibrillation/flutter are widely prevalent.
* Reported antiarrhythmic drug efficacy to restore & maintain sinus rhythm is 52% which is far from optimal.
* On the other hand, 5-year arrhythmia-free survival after catheter ablation was previously reported to be 63%.
* Therefore, there is a need for better characterization of the underlying atrial substrate, to improve treatment outcomes in terms of efficacy and safety

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years.
* Patients undergoing successful cardioversion (pharmacologic or electric) for atrial fibrillation/flutter, OR symptomatic patients with paroxysmal atrial fibrillation/flutter scheduled for trans-catheter ablation.
* Index cardioversion OR Index ablation procedure.

Exclusion Criteria:

* LA thrombus on TEE or CMR.
* Contraindications to CMR.
* Contraindications to Gd-based contrast.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Based on the previously reported antiarrhythmic drug efficacy of 52% in maintaining sinus rhythm:
  * For Wilcoxon-Mann-Whitney test for difference in 2 group means: assuming an alpha error probability of 0.05, a study power of 60-70%, and a 1:1 ratio of successful rhythm control vs atrial fibrillation/flutter recurrence, a total sample size of 86-106 would be needed (43-53 for each arm). [calculated by G*Power software v.3.1.9.7]
  * To be able to build multivariable logistic regression models including, e.g., 4-5 predictor variables, a reasonable sample size would be 80-100 patients.
  * Patient enrollment will continue until the projected sample size is satisfied or until 24 months have lapsed, whichever comes first.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Recurence in patient with AF or flutter after pharmacological or interventional rythm control | Baseline
  * Non-invasive rhythm control arm: Predictors of atrial fibrillation recurrence within 6 months of cardioversion or the need for ≥2 cardioversions in the 1st year after initial cardioversion.
  * Ablation arm: Predictors of success rate (acute and mid term) of ablation on multivariable logistic regression analysis.

SECONDARY OUTCOMES:
parameters for safe ablation | Baseline
  * Ablation arm: Predictors of esophageal thermal injury (ETI).
  * Arterial embolic events in both arms.

CONTACTS AND LOCATIONS:
Overall Officials: Salah EL-dein Sayed Ata, Professor of cardiology, Study Director — Assiut University
Locations (1):
- Assiut Univeristy Heart Hospital, Asyut, Egypt

REFERENCES:
- [Background] 1. Calkins H et al. Circ Arrhythm Electrophysiol. 2009